CLINICAL TRIAL: NCT04136457
Title: Proteome Remodelling and Dynamics in Human Skeletal Muscle: Effect of Training
Brief Title: Proteome Remodelling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MiDy
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Skeletal Muscle Physiology
MeSH Terms: interventions — Endurance Training; Resistance Training; High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endurance (Experimental): Endurance training
  Interventions: Other: Endurance training
- Resistance (Experimental): Resistance training
  Interventions: Other: Resistance training
- Sprint (Experimental): Sprint training
  Interventions: Other: Sprint training

INTERVENTIONS:
Other: Endurance training — Subjects perform a period of endurance training
  Arms: Endurance
Other: Resistance training — Subjects perform a period of resistance training
  Arms: Resistance
Other: Sprint training — Subjects perform a period of sprint training
  Arms: Sprint

SUMMARY:
The purpose of the project is to investigate the proteome signature dynamics and remodelling in human skeletal muscle induced by exercise training

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* VO2max > 55 mL/min/kgLM for men and > 50 for women (only applicable for endurance and sprint training interventions)
* BMI < 26

Exclusion Criteria:

* Chronic disease deemed by the medical doctor to pose a risk or to affect study outcomes
* smoking
* Use of prescription medicine deemed by the medical to affect study outcomes
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle proteome signature | Change from baseline at week 6 or 8 depending on the intervention
  Pathway enrichment analysis of the muscle proteome
Anabolic signaling | Change in anabolic signaling from rest to 1 hour following resistance exercise both at baseline and following 8 weeks of resistance training
  Western blotting of proteins related to anabolic signaling

SECONDARY OUTCOMES:
Skeletal muscle mitochondrial respiration | Change from baseline at week 6 following endurance and sprint training
  High resolution respirometry
Maximal oxygen consumption | Change from baseline at week 6 following endurance and sprint training
  VO2max during incremental exercise
Body composition | Change from baseline at week 6 or 8 depending on the intervention
  Lean and fat mass during dual X-ray absorptiometry
Myonuclei | Change from baseline at week 8 following resistance training
  Immunohistochemistry to determine number of myonuclei
Satellite cells | Change from baseline at week 8 following resistance training
  Immunohistochemistry to determine number of satellite cells
Fiber size | Change from baseline at week 8 following resistance training
  Immunohistochemistry to determine fiber size

OTHER OUTCOMES:
Skeletal muscle mitochondrial supercomplexes | Change from baseline at week 6 following endurance and sprint training
  Pathway enrichment analysis of mitochondrial supercomplexes

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kissow J, Jacobsen KJ, Jessen S, Thomsen LB, Quesada JP, Bangsbo J, Deshmukh AS, Hostrup M. Global Proteomics Reveals Distinct Muscle Adaptations to Menstrual Cycle Phase-Based Sprint Interval Training in Endurance-Trained Females. Mol Cell Proteomics. 2025 Oct;24(10):101053. doi: 10.1016/j.mcpro.2025.101053. Epub 2025 Aug 14. PMID 40818533